CLINICAL TRIAL: NCT05625932
Title: Prophylaxis of Venous Thromboembolic Disease With Low Molecular Weight (LMWH) (TINzaparin) in Patients With Metastatic Colorectal Cancer Who Start the First Line of Treatment.
Brief Title: TINzaparin Prophylaxis in Patients With Metastatic Colorectal Cancer
Acronym: PROTINCOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galician Research Group on Digestive Tumors (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GIT-PRo-2022-02; 2022-001534-11 (EudraCT Number)
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer Metastatic; Thromboembolism
Keywords: LMWH; Prophylaxis; Thromboembolic event; Colorectal cancer
MeSH Terms: conditions — Thromboembolism; Colorectal Neoplasms | interventions — Tinzaparin

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized, non-placebo controlled, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Those patients allocated in the control arm will receive no interventions related to VTE risk. No placebo will be administered to avoid discomfort of these patients who are already under treatment for their cancer.
- Experimental arm (Experimental): Those patients allocated to the experimental arm will receive prophylactic Tinzaparin at a fixed dose according to their weight:
  Patients < 80 kg will receive a fixed dose of 4500 IU daily. Patients between 80-100 kg will receive a fixed dose of 6000 IU daily. Patients > 100 kg will receive a fixed dose of 8000 IU daily.
  Accordingly, the effective dose of tinzaparin is estimated to be in the range of 56-90 IU/kg. Tinzaparin dose will be adjusted according to the dose levels specified above in patients who experience changes in body weight greater than 10% during treatment period.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — Patients < 80 kg will receive a fixed dose of 4500 IU daily. Patients between 80-100 kg will receive a fixed dose of 6000 IU daily. Patients > 100 kg will receive a fixed dose of 8000 IU daily.
  Other Names: Innohep
  Arms: Experimental arm

SUMMARY:
Patients with metastatic colorectal cancer (mCRC) who are scheduled to receive systemic cancer therapy have an increased risk for venous thromboembolic (VTE) events compared with the general population.

PROTINCOL is a randomized, open label, non placebo-controlled, low intervention, and phase III clinical trial that will recruit patients with mCRC. The study hypothesizes that prophylaxis with Tinzaparin could prevent the appearance of symptomatic and incidental VTE.

All patients will receive the first-line anticancer treatment deemed more appropriate according to the physician criteria. Enrolled patients are randomized in a 1:1 ratio (stratifying by BRAF/RAS, resection of primary tumor, and anti-angiogenic first-line treatment) to: control arm (no interventions related to VTE risk and no placebo) or experimental arm (prophylactic Tinzaparin at a fixed dose of 4500 IU/day in patients with up to 80kg, 6000 IU/day for those between 80-100 kg, or 8000 IU/day for those >100kg). Treatment is scheduled for a maximum period of 4 months. Treatment could be stopped earlier in case of unacceptable toxicity, patient consent withdrawal, physician criteria or end of study. Patients will undergo tumor and VTE assessments according to standard clinical practice.

The main objective of the study is to evaluate the efficacy of tinzaparin for the prevention of symptomatic or incidental VTE events. Secondary objectives include the associations between VTE events and tumor characteristics (i.e. laterality, RAS/BRAF mutations) or management (i.e. surgery or treatment with anti-angiogenic or anti-EGFR agents), cancer-specific survival outcomes, safety, the incidence of bleeding events, and patient-reported quality of life. The trial includes also a translational exploratory analysis to assess the predictive value of risk assessment models and genetic risk scores, their evolution through the study and microsatellite instability or other biomarkers.

DETAILED DESCRIPTION:
This research study is a prospective, randomized, open label (PROBE), non placebo-controlled, and phase III clinical trial; Investigator Initiated Study (IIS). The study has been considered a low-interventional clinical trial.

The trial will compare the efficacy and safety of tinzaparin with a watch and wait strategy for primary prophylaxis of symptomatic or incidental VTE in adult men and women, 18 years of age and older, with metastatic colorectal cancer who are scheduled to initiate systemic cancer therapy as a component of their standard of care anticancer regimen.

The study consists of 3 periods: a 4-week screening period, a 4 months treatment period and post-treatment follow-up period until the end of treatment (EOT) visit, scheduled 2 months after the last dose of tinzaparin or 6 months from the first dose of tinzaparin (whichever occurs latest). The duration of participation in the study for each subject is approximately 6 months. Further long-term phone follow-up to monitor for progression and survival could be carried out at the end of study. Tumor follow-up assessments will adhere to the standard clinical practice within each site.

All patients will receive the first-line anticancer treatment deemed more appropriate according to the physician criteria and current guideline recommendations. Patients in both groups will receive supportive care as per local practice. No formal recommendations will be issued by the study protocol regarding cancer treatment and supportive care, but the drugs used will be recorded in the clinical report form. Constitutive use of anticoagulant drugs will be prohibited during the treatment period.

Enrolled patients are randomized in a 1:1 ratio to the control arm, or the experimental arm:

Control arm: A watch and wait strategy will be used. There is no placebo. Since no reference treatment is available for long-term VTE prophylaxis in patients with cancer, patients in the control group will not receive VTE prophylaxis outside the hospital and will receive anticancer treatment and supportive care as per local practice. No formal recommendations will be issued by the study protocol regarding cancer treatment and supportive care, but the drugs used will be recorded in the clinical report form (CRF). Patients in the control group will receive antithrombotic prophylaxis as per local practice during hospitalizations. Any use of LMWH will be recorded in the CRF.

Experimental arm: Patients will receive prophylaxis tinzaparin at a fixed dose daily for 4 months.

The primary objective is to evaluate the efficacy of 4-months prophylaxis with tinzaparin for the prevention of symptomatic or incidental VTE events. Secondary efficacy objectives include the VTE incidence in specific subpopulations (stratification according to the laterality of the primary tumor, first-line treatment with anti-EGFR or antiangiogenics, and mutational status).

Safety of tinzaparin will be evaluated by means of relevant adverse events, incidence of bleedings according to International Society of Thrombosis and Hemostasis (ISTH) criteria, and patient-reported quality of life. Bleeding events will be evaluated locally by the investigator and centrally by a blinded committee.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with age ≥ 18 years.
2. Written informed consent.
3. Patients with a histologically confirmed diagnosis of stage IV colon or rectal adenocarcinoma (mCRC).
4. Locally assessed BRAF and RAS genomic alterations available during screening.
5. Beginning of the first line of treatment for metastatic disease with chemotherapy +/- targeted therapy (i.e. antiangiogenic, anti-EGFR, encorafenib-cetuximab doublet) or immunotherapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Life expectancy >6 months.

Exclusion Criteria:

1. Contraindication to tinzaparin, or other heparins:

   1. Allergy (or hypersensitivity) to heparin, tinzaparin, other LMWHs, or pork products.
   2. History or presence of heparin-induced (type II) thrombocytopenia.
   3. Have or have had an epidural catheter or a traumatic spinal puncture within the previous 7 days.
2. Prothrombin time (PT) (International normalized ratio [INR] >1.5 for any reason) or aPTT >2 times control value.
3. Active major bleeding or conditions predisposing to major bleeding. a major bleeding is defined as one that meets one of the following three criteria:

   1. occurring in a critical area or organ (for example, intracranial, intra-spinal, intraocular, retroperitoneal, intra-articular or pericardial, intrauterine or intramuscular with compartment syndrome),
   2. causing a decrease in hemoglobin levels of 2 g/l (1.24 mmol/l) or more, or that requires a transfusion of two or more units of whole blood or packed red blood cells.
4. Lesions or conditions at increased risk of clinically significant bleeding, including:

   1. Previously diagnosed/treated VTE ≤ 28 days prior to randomization.
   2. Active ulcer disease.
   3. Diagnosed cerebral metastases.
   4. Stroke within the prior 6 months.
   5. History of central nervous system (CNS) or intraocular bleeding.
5. Requirement of other anticoagulant therapy, dual antiplatelet therapy, daily non-steroidal anti-inflammatory drugs, or other medications known to increase the risk of bleeding.

   Note: A daily dose of ≤100 mg of aspirin and single agent clopidogrel are permitted
6. Acute or chronic renal insufficiency with Creatinine clearance < 30 ml / min.
7. Platelet count < 80.000 /ml at the time of inclusion.
8. Severe liver insufficiency as defined by clinical manifestations of ascites, cirrhosis, encephalopathy and/or jaundice and/or biochemical abnormalities in liver function tests including:

   1. elevated levels of total bilirubin (> 2 times the upper limit normal [ULN]),
   2. elevated liver transaminases (> 2 times the ULN; > 5 in case of hepatic metastasis).
9. Participating in another study of an investigational agent at the time of enrollment. Note: Use of an experimental regimen of an approved product is not cause for exclusion.
10. Patients who weigh < 50 Kg.
11. Women of childbearing potential (WOCBP), must provide a negative serum or urine pregnancy test at screening. Women breastfeeding are not eligible.

    Note: A pregnancy test is performed on WOCBP as per standard of care for patients undergoing anticancer treatments.
12. Any underlying medical or psychiatric disorder, which, in the opinion of the investigator, makes the administration of tinzaparin unsafe or interferes with the informed consent process or trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence of any VTE | Throughout the study period, approximately 6 months per patient
  The primary efficacy endpoint is the cumulative incidence (percentage of patients) of any VTE event including:
  Symptomatic non-fatal pulmonary thromboembolism (PE). Symptomatic lower-limb deep vein thromboembolism (sllDVT). Symptomatic upper extremity deep vein thromboembolism (sueDVT). Incidentally diagnosed PE or proximal DVT. Symptomatic central venous catheter thromboembolism. Incidentally visceral vein thrombosis (iVVT). Symptomatic visceral vein thrombosis (sVVT). VTE-related deaths

SECONDARY OUTCOMES:
Incidence of symptomatic non-fatal PE | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of sllDVT | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of sueDVT | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of incidentally diagnosed PE or proximal DVT | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of symptomatic central venous catheter thromboembolism | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of iVVT | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of sVVT | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of VTE-related deaths | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing the event during the observation period (6 months)
Incidence of confirmed VTE events in BRAF/RAS mutated patients | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients with BRAF / RAS tumor genomic mutations vs native BRAF / RAS tumors.
Incidence of confirmed VTE events in resected or not resected patients | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients with primary tumor resection vs not resection.
Incidence of confirmed VTE events in patients with antiangiogenic therapy | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients on antiangiogenic treatment
Incidence of confirmed VTE events in patients with anti-EGFR therapy | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients on anti-EGFR treatment
Incidence of confirmed VTE events in patients according to tumor laterality | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients with right-side / transverse primary tumor vs left-side primary tumor.
Incidence of confirmed VTE events in patients according to progression (PD) | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients with PD according to usual clinical practice determined by the treating physician during treatment with tinzaparin
Incidence of confirmed VTE events in patients according genetic risk scores | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients according to their genetic risk score
Incidence of confirmed VTE events in patients according to blood type | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing confirmed VTE events in patients according to their blood type
Incidence of arterial thromboembolic events (ATE) | Throughout the study period, approximately 6 months per patient
  Percentage of patients experiencing ATE
Thrombosis-free survival (TFS) | Throughout the study period, approximately 6 months per patient
  Defined as the time elapsed from the first dose of study treatment to the diagnosis of thrombotic event, or death from any cause, whichever occurs first
Event-free survival (EFS) | Throughout the study period, approximately 6 months per patient
  Events are defined as the endpoint of mortality, major bleeding and VTE. EFS is defined as the time elapsed from the first dose of study treatment to the diagnosis of VTE event, major bleeding event, or death by any cause, whichever occurs first
Progression-free survival (PFS) | Throughout the study period, approximately 6 months per patient
  Defined as the time elapsed from the first dose of study treatment to progression determined by the treating physician according to local standard clinical practice, or death from any cause, whichever occurs first
Overall survival (OS) | Throughout the study period, approximately 6 months per patient
  Defined as the time elapsed from the first dose of study treatment until death from any cause
Mortality rate | Throughout the study period, approximately 2 years
  Percentage of patients who died through the study
Incidence of relevant adverse events (AE) | Throughout the study period, approximately 2 years
  Percentage of patients who experience grade 3-5 according to CTCAE version 5.0
Incidence of treatment-related AEs (TRAEs) | Throughout the study period, approximately 2 years
  Percentage of patients who experience TRAEs
Incidence of major bleeding (MB) events | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experience MB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment
Incidence of Clinically relevant non-major bleeding (CRNMB) | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experience CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment
Quality of life score | Throughout the study period, approximately 6 months per patient
  Patients reported outcomes through the EORTC quality of life questionnaire (QLQ)-C30 questionnaire. QLQ-C30 scale is a 28 items that are scored on a 4-point response scale. All scale scores are linearly converted to range from 0 to 100. For the functioning scales and global QOL higher scores indicate better functioning.
Incidence of bleeding events in BRAF/RAS mutated patients | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported according to BRAF/RAS mutational statu
Incidence of bleeding events according to surgery | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported according to previous surgery of the primary tumor
Incidence of bleeding events according to antiangiogenic therapy | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported according to first-line antiangiogenic agents treatment
Incidence of bleeding events according to anti-EGFR therapy | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported according to first-line anti-EGFR treatment
Incidence of bleeding events according to tumor laterality | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported in patients with right-sided or transversal vs. left-sided primary tumor
Incidence of bleeding events according to genetic risk | Throughout the study period, approximately 6 months per patient
  Percentage of patients who experienced a MB or CRNMB according to ISTH criteria throughout the study period and up to month 2 of end of tinzaparin treatment. Results will be reported in patients according to their genetic risk score

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Salgado, M.D. Ph.D., Study Chair — Complexo Hospitalario Universitario de Ourense (Galicia); Andrés Muñoz, M.D. Ph.D., Study Chair — Hospital Universitario Gregorio Marañón (Madrid)
Locations (35):
- Spain (35):
  - Hospital Clínico Universitario de Santiago CHUS, Santiago de Compostela, A Coruña
  - Hospital Público Verge dels Lliris, Alcoy, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - ICO (Institut Català d'Oncologia) de Badalona, Badalona, Barcelona
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Consorcio Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Univ. de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Príncipe de Asturias (HUPA) de Alcalá de Henares, Alcalá de Henares, Madrid
  - Hospital Universitario De Móstoles, Móstoles, Madrid
  - Hospital Infanta Cristina (Parla), Parla, Madrid
  - Hospital Universitario Infanta Elena, Valdemoro, Madrid
  - Hospital Costa del Sol de Marbella, Marbella, Málaga
  - Hospital Obispo Polanco De Teruel, Teruel, Terul
  - Complejo Hospitalario Universitario de A Coruña (CHUAC), A Coruña
  - Centro Oncológico de Galicia (A coruña), A Coruña
  - Complejo Hospitalario Universitario de Ferrol ( Arquitecto Macide), A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Virgen de la Luz de Cuenca, Cuenca
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario Universitario De Ourense, Ourense
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra
  - Complejo Asistencial Universitario De Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital General Universitario de Toledo, Toledo
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Ribera Povisa, Vigo
  - Complejo Hospitalario Universitario de Vigo (Álvaro Cunqueiro), Vigo
  - Complejo Asistencial de Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No
Anonymized individual participant data (IPD) may be available upon request if it is within the same scope approved by the participants when they gave their written informed consent to participate

REFERENCES:
- [Derived] Salgado M, de la Camara-Gomez J, Garcia-Escobar I, Alvarez-Llosa RC, Gonzalez-Villarroel P, Garay DF, Pampols-Felip M, Guillot-Morales M, Pelegrin-Mateo FJ, Jimenez-Orozco E, Sastre J, de Castro EM, Coma E, Bouzas LP, Ferrer-Perez AI, Momprade-Olive E, Cousillas-Castineiras A, Covela-Rua M, Rojas M, Querol R, Diaz LR, Merino M, Gil M, Sanchez-Canovas M, Elias T, Marrupe-Gonzalez D, Sanchez-Gil B, Carmona-Campos M, Garcia-Ferron M, Soria JM, Munoz A. Tinzaparin for the prevention of thromboembolic events in ambulatory patients with metastatic colorectal cancer receiving first line treatment: a randomised, clinical trial design. BMC Cancer. 2025 Nov 17;25(1):1773. doi: 10.1186/s12885-025-14620-z. PMID 41249955